CLINICAL TRIAL: NCT02511535
Title: TBE (Tick-borne Encephalitis ) Vaccination in Allergic Patients
Brief Title: TBE (Tick-borne Encephalitis) Vaccination in Allergic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Ursula Wiedermann, Univ.-Prof. Dr. Ursula Wiedermann, MD, PhD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TBE_1.1
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Vaccine Responsiveness in Allergy; Vaccine Responsiveness During Allergy De-sensitization Treatment
MeSH Terms: interventions — FSME-IMMUN vaccine; Dimenhydrinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Allergic patients (Experimental): Allergic patients receive TBE booster vaccination
  Interventions: Biological: TBE booster vaccination
- Allergic patients with de-sensitization treatment (Experimental): Allergic patients with de-sensitization treatment receive TBE booster vaccination
  Interventions: Biological: TBE booster vaccination
- Healthy controls (Active Comparator): Healthy controls receive TBE booster vaccination
  Interventions: Biological: TBE booster vaccination

INTERVENTIONS:
Biological: TBE booster vaccination
  Other Names: Vaccine: FSME-Immun® (Fruehsommer-Meningoencephalitis); One dose (0.5 ml) contains:; 2.4 micrograms Tick-Borne Encephalitis Virus ( strain Neudoerfl),; adsorbed on aluminium oxide, hydrated (0.35 milligrams Al3+); Manufacturer: Baxter Innovations GmbH

SUMMARY:
Allergic patients especially those undergoing de-sensitization treatment have an altered immune responsiveness. The investigators aim to find out whether this influences immune responses to primary and booster vaccinations.

DETAILED DESCRIPTION:
Allergic patients generally have an altered immunologic profile (Th2 bias), and allergic individuals undergoing de-sensitization treatment display an increased production of immune suppressive cytokines. The investigators measure humoral and cellular immune responses to routine vaccination (Tick-borne Encephalitis [TBE] booster) in allergic patients with and without de-sensitization treatment to determine whether allergy negatively influences vaccine induced immune responses and protection.

ELIGIBILITY:
Inclusion Criteria:

* completed primary TBE immunization + at least one booster immunization
* adults of both sexes between 18 and 60 years of age
* willingness to sign written informed consent form

Exclusion Criteria:

* age < 18 and > 60 years
* prior TBE infection
* Hepatitis A vaccination
* pregnancy and breast feeding
* acute infection on day of inclusion (day 0), body temperature >37,9°C
* concomitant medications: systemic cortisone therapy, chemotherapy, immunosuppressive therapy 4 weeks prior to or during study
* administration of other vaccines 4 weeks before/after TBE vaccination
* planned surgery within 2 weeks before/after TBE vaccination
* Start of de-sensitization and the first 4 weeks of allergen dose escalation
* any contraindication to administration of FSME-Immun® vaccine according to manufacturer's instructions
* history of malignant disease within the last 5 years
* autoimmune diseases
* drug addictions
* plasma donors
* receipt of blood transfusions or immuno globulins within 3 month before study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann, MD, PhD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Institute of Specific Prophylaxis and Tropical Medicine, Vienna, Austria

REFERENCES:
- [Derived] Garner-Spitzer E, Seidl-Friedrich C, Zwazl I, Hofer M, Kinaciyan T, Jarisch R, Stiasny K, Zlabinger GJ, Kundi M, Wiedermann U. Allergic patients with and without allergen-specific immunotherapy mount protective immune responses to tick-borne encephalitis vaccination in absence of enhanced side effects or propagation of their Th2 bias. Vaccine. 2018 May 11;36(20):2816-2824. doi: 10.1016/j.vaccine.2018.03.076. Epub 2018 Apr 16. PMID 29673942

RESULTS

PARTICIPANT FLOW:
Groups:
- Allergic Patients: Allergic patients receive TBE booster vaccination
  TBE booster vaccination
- Allergic Patients With De-sensitization Treatment: Allergic patients with de-sensitization treatment receive TBE booster vaccination
  TBE booster vaccination
- Healthy Controls: Healthy controls receive TBE booster vaccination
  TBE booster vaccination
Period: Overall Study
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
Started | 49 | 21 | 49
Completed | 49 | 21 | 49
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls | Total
Number analyzed (Participants) | 49 | 21 | 49 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 21 | 49 | 119
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 12 | 30 | 72
  Male | 19 | 9 | 19 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 21 | 49 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 49 | 21 | 49 | 119

OUTCOME MEASURES:

1. Primary Outcome: Humoral TBE Immunity
Description: Geometric mean titers of TBE specific neutralizing Abs
Time Frame: one month after booster vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
Number analyzed (Participants) | 49 | 21 | 49
titer | 317.90 [238.70 to 423.30] | 250.10 [143.90 to 434.40] | 282.20 [210.60 to 378.20]

2. Secondary Outcome: Cellular Immune Response - Cytokine Production
Description: cytokine production of antigen-specifically re-stimulated PMBC, IL-2 (interleukin 2) IFN g (interferon gamma) IL-10 (interleukin 10) IL-5 (interleukin 5)
Time Frame: before (day 0) and 1week after booster vaccination
Population: the missing cytokine concentrations were not used for calculation because of invalid positive controls (due to poor PBMC [peripheral blood mononuclear cell] viability)
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
Number analyzed (Participants) | 49 | 21 | 49
pg/ml
  IFNg before vaccination | 37.85 [25.86 to 55.39] | 42.54 [23.36 to 77.49] | 38.91 [25.13 to 59.01]
  IFNg 1 week post vacc: number analyzed (Participants) | 48 | 21 | 47
  IFNg 1 week post vacc | 54.19 [37.61 to 78.08] | 59.45 [32.67 to 108.17] | 77.27 [52.26 to 114.25]
  IL-10 before vaccination | 35.21 [25.90 to 47.86] | 38.86 [23.75 to 63.58] | 30.28 [21.15 to 43.37]
  IL-10 one week post vacc: number analyzed (Participants) | 48 | 21 | 49
  IL-10 one week post vacc | 48.90 [36.60 to 65.33] | 52.13 [37.00 to 73.44] | 52.28 [36.47 to 74.95]
  IL-2 before vaccination | 52.62 [36.54 to 75.78] | 35.41 [21.25 to 59.02] | 37.20 [24.43 to 56.64]
  IL-2 one week post vacc: number analyzed (Participants) | 48 | 21 | 49
  IL-2 one week post vacc | 53.80 [37.03 to 78.18] | 37.11 [24.44 to 56.34] | 51.07 [34.57 to 75.44]
  IL-5 before vaccination | 2.08 [1.81 to 2.40] | 1.85 [1.85 to 1.85] | 2.04 [1.87 to 2.23]
  IL-5 one week post vaccination: number analyzed (Participants) | 48 | 21 | 49
  IL-5 one week post vaccination | 2.96 [2.32 to 3.77] | 1.87 [1.84 to 1.90] | 2.85 [2.23 to 3.64]

3. Secondary Outcome: Cellular Immune Response - Lymphocyte Subpopulations
Description: analyses of naive, memory and regulatory sub-populations of B- and T-lymphocytes
Time Frame: before (day 0) and 1week after booster vaccination
Measure: Mean (95% Confidence Interval); unit: percent of total lymphocytes
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
Number analyzed (Participants) | 49 | 21 | 49
percent of total lymphocytes
  T cells (CD3 +) at day 0 | 69.3 [66.9 to 71.8] | 73.7 [70.9 to 76.5] | 68.2 [65.5 to 71.0]
  T cells (CD3 +) 1 week after booster vaccination | 68.7 [66.1 to 71.2] | 74.7 [72.4 to 77.1] | 70.6 [68.3 to 72.9]
  B cells (CD19 +) at day 0 | 7.63 [6.67 to 8.57] | 7.01 [6.04 to 7.98] | 7.11 [6.34 to 7.89]
  B cells (CD19 +) 1 week after booster vaccination | 7.22 [6.33 to 8.11] | 6.34 [5.34 to 7.34] | 6.39 [5.78 to 7.01]
  T helper cells (CD4 +) at day 0 | 42.3 [39.9 to 44.6] | 49.1 [45.5 to 52.4] | 41.6 [38.7 to 44.4]
  T helper cells (CD4 +) 1 week after booster | 42.7 [40.4 to 45.0] | 50.5 [47.6 to 53.4] | 43.0 [40.1 to 45.8]
  cytotoxic T cells (CD8 +) at day 0 | 21.5 [19.8 to 23.3] | 20.3 [17.0 to 23.4] | 20.6 [18.4 to 22.8]
  cytotoxic T cells (CD8 +) 1 week after booster | 20.9 [19.3 to 22.6] | 20.7 [17.5 to 23.8] | 21.2 [19.0 to 23.3]
  Tregs (CD4+ FOXP3+) at day 0 | 4.65 [4.20 to 5.13] | 5.36 [4.61 to 6.16] | 4.49 [4.10 to 4.89]
  Tregs (CD4+ FOXP3+) 1 week after booster | 4.54 [4.10 to 5.01] | 5.60 [4.93 to 6.30] | 4.21 [3.84 to 4.60]

4. Secondary Outcome: TBE Titer Course
Description: Fold Change in TBE Specific Neutralizing Antibodies from day 0 (before booster) and one week, one month and 6 months after booster vaccination
Time Frame: before (day 0) until 6 months after booster vaccination
Measure: Mean (95% Confidence Interval); unit: fold change from d0 (before booster)
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
Number analyzed (Participants) | 49 | 21 | 49
fold change from d0 (before booster)
  fold change 1 week after booster | 1.46 [1.23 to 1.73] | 1.80 [1.36 to 2.37] | 1.79 [1.50 to 2.14]
  fold change 4 weeks after booster | 3.02 [2.43 to 3.77] | 3.01 [2.05 to 4.41] | 2.56 [2.09 to 3.13]
  fold change 6 month after booster | 1.95 [1.54 to 2.46] | 2.53 [1.81 to 3.54] | 1.79 [1.41 to 2.29]

ADVERSE EVENTS:
Arm/Group | Allergic Patients | Allergic Patients With De-sensitization Treatment | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/21 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/21 | 0/49
Other Adverse Events (participants affected / at risk) | 23/49 | 12/21 | 27/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Allergic Patients (N=49) | Allergic Patients With De-sensitization Treatment (N=21) | Healthy Controls (N=49)
vaccine reactogenicity (Skin and subcutaneous tissue disorders) | 23 | 12 | 27 — local reactions to TBE vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes